CLINICAL TRIAL: NCT00137605
Title: A Pilot Study Assessing the Efficacy of Pneumococcal Vaccine in HIV Patients: Delayed Versus Immediate Immunization
Brief Title: Early Versus Delayed Pneumococcal Vaccination in HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CIHR Canadian HIV Trials Network (Network)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CTN 147; Control # 078760; File # 9427-C1574-34C
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Pneumococcal Infections
Keywords: HIV; HIV Infections
MeSH Terms: conditions — Pneumococcal Infections; HIV Infections | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

ARMS (4):
- Pneumovax/immediate (Experimental)
  Interventions: Biological: Pneumovax
- Pneumovax/delayed (Experimental)
  Interventions: Biological: Pneumovax
- Prevnar/immediate (Experimental)
  Interventions: Biological: Prevnar
- Prevnar/delayed (Experimental)
  Interventions: Biological: Prevnar

INTERVENTIONS:
Biological: Pneumovax
  Arms: Pneumovax/delayed; Pneumovax/immediate
Biological: Prevnar
  Arms: Prevnar/delayed; Prevnar/immediate

SUMMARY:
The purpose of this study is to determine whether people who are HIV-positive respond better to a vaccine for pneumonia-related disease when they are immunized immediately, or when immunization is delayed until the immune system has improved to a certain level. The study will also compare the effectiveness of polysaccharide and heptavalent vaccines.

DETAILED DESCRIPTION:
A multicentre, randomized controlled trial using a two factorial design. Eighty patients will be randomly assigned to receive either Pneumovax (or Pneumo23 according to standard use at site) or heptavalent pneumococcal conjugate vaccine (Prevnar) prior to reconstitution of the immune system or will have immunization delayed until their CD4 count is greater than 200 cells/mm3 after the introduction of antiretroviral therapy. Randomization will be stratified by study centre. Variable block sizes will be used to try to prevent study personnel from guessing the next allocation. Random allocation lists will be generated by computer.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Between 18 and 65 years of age
* Have a CD4 cell count below 200 cells/mm3
* Willing to begin/change antiretroviral therapy
* Willing and able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Have had previous pneumococcal vaccination
* Have had occurrence of pneumococcal infection (brain, blood or lung infections) in past 5 years
* Have hypersensitivity to components of either vaccine
* Have acute feverish illness at the time of vaccination
* Have had splenectomy (removal of the spleen)
* Have received treatment with IVIG within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of serotypes to which a response is found
A response is defined as a doubling in antibody titer at 1 month compared to baseline.

SECONDARY OUTCOMES:
Antibody response at 6 months and one year
Changes in viral load 3 months post immunization
Adverse events
Overall incidence of invasive pneumococcal disease
Incidence of invasive pneumococcal disease between vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Walter Schlech, MD, Principal Investigator — Victoria General Hospital
Locations (14):
- Canada (14):
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Downtown IDC, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Moncton Hospital, Windsor, New Brunswick
  - Victoria General, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Sunnybrook, Toronto, Ontario
  - Toronto General, Toronto, Ontario
  - Metropolitan Hospital, Windsor, Ontario
  - Montreal Chest/Royal-Victoria, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Laval, Ste-Foy, Quebec

REFERENCES:
- [Result] Slayter KL, Singer J, Lee TC, Kayhty H, Schlech WF. Immunization against pneumococcal disease in HIV-infected patients: conjugate versus polysaccharide vaccine before or after reconstitution of the immune system (CTN-147). Int J STD AIDS. 2013 Mar;24(3):227-31. doi: 10.1177/0956462412472450. Epub 2013 May 6. PMID 23535358
- [Derived] Kimby E, Schar S, Pirosa MC, Vanazzi A, Mey UM, Rauch D, Wahlin BE, Hitz F, Hernberg M, Johansson AS, de Nully Brown P, Hagberg H, Ferreri AJM, Krasniqi F, Voegeli M, Novak U, Zander T, Bersvendsen H, Mamot C, Mingrone W, Stathis A, Dirnhofer S, Hayoz S, Ostenstad B, Zucca E. Six-month rituximab-lenalidomide regimen in advanced untreated follicular lymphoma: SAKK 35/10 trial 10-year update. Blood Adv. 2025 Apr 8;9(7):1712-1719. doi: 10.1182/bloodadvances.2024014840. PMID 39883948